CLINICAL TRIAL: NCT06352177
Title: Efficacy of a Novel Digital Therapeutic Lifestyle Intervention Program for Patients With MASLD
Brief Title: Digital Therapeutic Lifestyle Intervention Program for Patients With MASLD
Acronym: ENLIGHTEN
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal investigator left the institution and study was never funded
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Stephanie Patton, Compliance Specialist, Penn State Health, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: protocol-1
Record Dates: First submitted 2024-02-08; First posted 2024-04-08 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: NASH; NASH - Nonalcoholic Steatohepatitis; Liver Diseases
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Liver Diseases

STUDY DESIGN:
Intervention Model Description: 2:1 randomization
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention): Participants in this group will receive counseling about best MASLD clinical practices in accordance with AASLD and ACSM practice guidelines Because in-office hepatology counseling for lifestyle intervention occurs every 12-24 wks,standard counseling will occur at each in-person visit. Mediterranean-informed, hypocaloric dietary counseling will be provided by a study investigator, with specific instructions to limit carbohydrates and saturated fat and enrich dietary intake with high fiber and unsaturated fats. Physical activity goals of 150 min/wk. of moderate intensity of 75 min/wk. of vigorous intensity activity will be suggested. To reinforce this education and promote self-monitoring, participants in this group will also receive a digital scale and fitness activity tracker.
- Intervention (Experimental): This commercially available program (Noom Weight) promotes clinically significant body weight loss and behavior change in multiple populations including our pilot study in individuals with MASLD. The program is delivered through a smartphone application and includes self-monitoring and feedback features for diet, physical activity, and body weight, as well as digital access to a 1:1 behavior change coach, a support group facilitated by a health coach, and a curriculum delivered via daily articles focused on nutrition, physical activity, and sustainable behavioral change.
  Interventions: Other: Noom Weight Application

INTERVENTIONS:
Other: Noom Weight Application — This commercially available program (Noom Weight) promotes clinically significant body weight loss and behavior change in multiple populations. The program is delivered through a smartphone application and includes self-monitoring and feedback features for diet, physical activity, and body weight, as well as digital access to a 1:1 behavior change coach, a support group facilitated by a health coach, and a curriculum delivered via daily articles focused on nutrition, physical activity, and sustainable behavioral change.
  Other Names: NW
  Arms: Intervention

SUMMARY:
The ENLIGHTEN study that will evaluate the efficacy of a novel DTx lifestyle intervention in participants with non-cirrhotic MASH. People who have MASH, the progressive subtype of MASLD, have the highest risk for liver disease progression and poor outcomes, including cirrhosis and hepatocellular carcinoma, and greater overall mortality. Thus, these participants are expected to experience the greatest benefit from treatment.

This is a randomized, controlled trial comparing DTx lifestyle intervention in participants with non-cirrhotic MASH to standard clinical care. The study includes a screening period (up to 2 wks.) followed by randomization, 52-wk treatment period and 12-wk follow-up period (total duration up to 64 wks.).

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years at the time of signing informed consent
2. MASH defined by any of the following within 12-months prior to SV (V1):

   1. Liver biopsy with definitive MASH with NAS >4 with >1 in each component (i.e., steatosis, lobular inflammation, ballooning) or;
   2. Imaging study (e.g., ultrasound) with hepatic steatosis and one of the following:

   i) FIB-4 >1.3 or; ii) ELF test >7.7 or; iii) VCTE measured liver stiffness >8kPa or FAST score >0.35 or; iv) MRE measured liver stiffness >2.55kPa or MAST score >0.165
3. Possession of a smartphone (iPhone6s or newer with iOS version 15.6 or above; Android device with Android version 6 or above)
4. If participants are on GLP1-RA or other regulatory agency approved anti-obesity medication (e.g., orlistat, buproprion/naltrexone, phentermine-topiramate, phentermine, loreaserin), the medication dose must be stable (no change in dose) for the 3 mos. before SV.
5. Stable body weight for 3 mos. before screening visit defined as <5% weight loss or weight gain

Exclusion Criteria:

1. Recent (within 3 mos. of SV) participation in lifestyle intervention program or use of supplements marked for weight loss or appetite.
2. Plans to undergo bariatric surgery or initiate anti-obesity medication.
3. History of cirrhosis and/or hepatic decompensation (e.g., ascites, encephalopathy, variceal bleeding)
4. Liver disease of other etiologies (e.g., viral hepatitis), including liver transplantation
5. History of excessive alcohol consumption defined by self-report (men >30g/d or women >20g/d), AUDIT-C >4 or PETH > 20ug/L
6. History of malignancy within last 5 yrs., excluding successful treatment of non-melanoma skin cancer
7. Participant in any clinical trial or use of drugs under investigation for treatment of MASH within 3 mos. of SV
8. History of type 1 diabetes or uncontrolled type 2 diabetes (A1c >9.5% or changes in diabetes medication doses within 3 mos. of SV)
9. Recent (within 3 mos. of SV) initiation or change in dose of medications used to treat MASH (e.g., vitamin E, pioglitazone)
10. Recent (within 3 mos. of SV) use of drugs associated with the development of steatotic liver disease (e.g., methotrexate, tamoxifen)
11. Known or suspected history of drug abuse within the last 2 years prior to SV at the discretion of study investigator
12. Vulnerable participants (e.g., protected adults under guardianship or committed to an institution by governmental or judicial order)
13. Participants who cannot communicate with the study investigators or use digital technology reliably
14. Severe medical comorbidities that may hinder study participation at the discretion of study investigator
15. Current pregnancy or plans to become pregnant during the study period

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2030-01-01 (Estimated); Study Completion 2030-04-01 (Estimated)

PRIMARY OUTCOMES:
Clinically significant liver fat loss | 16 weeks
  Proportion of participants achieving >30% relative reduction in MRI-PDFF after Wk. 16.

SECONDARY OUTCOMES:
Sustained clinically significant body weight loss | 16 weeks
  Proportion of participants achieving >5% body weight loss after Wk. 16.
Sustained clinically significant body weight loss | 52 weeks
  Proportion of participants achieving >5% body weight loss after Wk. 52
Liver fat and liver stiffness using imaging analysis | 16 weeks
  • VCTE will assess change in liver fat and stiffness at Wks. 16
Liver fat and liver stiffness using imaging analysis | 16 weeks
  • MRI-PDFF will assess change in liver fat at Wks. 16
Liver fat and liver stiffness using imaging analysis | 16 weeks
  • MRE will assess change in liver stiffness at Wks. 16
Liver fat and liver stiffness using imaging analysis | 52 weeks
  VCTE will assess change in liver fat and stiffness at Wks. 52.
Liver fat and liver stiffness using imaging analysis | 52 weeks
  • MRI-PDFF will assess change in liver fat at Wks. 52.
Liver fat and liver stiffness using imaging analysis | 52 weeks
  • MRE will assess change in liver stiffness at Wks. 52
Clinically meaningful improvement in liver fat and stiffness | 16 weeks
  • Proportion of participants with >26% relative reduction in VCTE-measured liver stiffness (kPA) after Wks. 16
Clinically meaningful improvement in liver fat and stiffness | 16 weeks
  • Proportion of participants with >30% relative reduction in MRI-PDFF after Wk. 16
Clinically meaningful improvement in liver fat and stiffness | 16 weeks
  • Proportion of participants with >15% decrease in MRE-measured liver stiffness (kPA) after Wks. 16
Clinically meaningful improvement in liver fat and stiffness | 52 weeks
  • Proportion of participants with >26% relative reduction in VCTE-measured liver stiffness (kPA) after Wks. 52
Clinically meaningful improvement in liver fat and stiffness | 52 weeks
  • Proportion of participants with >30% relative reduction in MRI-PDFF after Wk. 52
Clinically meaningful improvement in liver fat and stiffness | 52 weeks
  • Proportion of participants with >15% decrease in MRE-measured liver stiffness (kPA) after Wks. 52
Circulating biomarkers of hepatic injury | 16 Weeks
  • Change in ALT after Wks. 16
Circulating biomarkers of hepatic injury | 16 Weeks
  • Proportion of participants with >17 IU/L decrease in ALT after Wks. 16
Circulating biomarkers of hepatic injury | 16 Weeks
  • Change in AST after Wks. 16
Circulating biomarkers of hepatic injury | 16 Weeks
  • Change in CK-18 after Wks. 16
Circulating biomarkers of hepatic injury | 16 Weeks
  • Change in GGT after Wks. 16
Circulating biomarkers of hepatic injury | 16 Weeks
  • Change in NASH Fibrotic Index after Wks. 16
Circulating biomarkers of hepatic injury | 16 Weeks
  • Proportion of participants with >17 IU/L decrease in ALT after Wks. 16.
Circulating biomarkers of hepatic injury | 52 weeks
  • Change in ALT after Wks. 52
Circulating biomarkers of hepatic injury | 52 weeks
  • Change in AST after Wks. 52
Circulating biomarkers of hepatic injury | 52 weeks
  • Change in CK-18 after Wks. 52
Circulating biomarkers of hepatic injury | 52 weeks
  • Change in GGT after Wks. 48.
Circulating biomarkers of hepatic injury | 52 weeks
  • Change in NASH Fibrotic Index after Wks. 52.
Circulating biomarkers of hepatic injury | 52 weeks
  • Proportion of participants with >17 IU/L decrease in ALT after Wks. 52
Circulating biomarkers of liver fibrosis and fibrogenesis | 16 Weeks
  • Change in Enhanced Liver Fibrosis (ELF) score after Wks. 16
Circulating biomarkers of liver fibrosis and fibrogenesis | 16 Weeks
  • Change in Fibrosis-4 index (FIB-4) after Wks. 16
Circulating biomarkers of liver fibrosis and fibrogenesis | 16 Weeks
  • Change in PRO-C3 after Wks. 16
Circulating biomarkers of liver fibrosis and fibrogenesis | 52 weeks
  • Change in Enhanced Liver Fibrosis (ELF) score after Wks. 52
Circulating biomarkers of liver fibrosis and fibrogenesis | 52 weeks
  • Change in Fibrosis-4 index (FIB-4) after Wks. 52
Circulating biomarkers of liver fibrosis and fibrogenesis | 52 weeks
  • Change in PRO-C3 after Wks. 52

IPD SHARING:
Plan to Share IPD: Yes
For this project, we anticipate data from 120 participants enrolled into the ENLIGHTEN study. There will be ten data collection points over the study duration. We will collect demographic, clinical, quality of life and outcomes information. Data will be converted to SAS and csv formats for analysis and sharing. To protect research participant personal identifying information (PII) and protected health information (PHI), all data will be de-identified prior to receipt by the repository and sharing in accordance with guidance provided for Limited Data Sets and Data Use Agreements section of NIH HIPAA Privacy Rule summary.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: We agree to deposit all data into the repository as soon as possible but no later than within one year of the completion of the funded project period for the parent award or upon acceptance of the main outcome data for publication. The data shared will be archived and available on the platform for request by researchers for a minimum of 10 years after contribution. Data will be made accessible no later than the time of our associated publication or the end of the grant period (whichever comes first).
Access Criteria: We will make the data available via the Vivli platform. Vivli is a non-profit clinical research data sharing platform that has been created to meet the needs of researchers who use and produce clinical research data worldwide. Using the Vivli platform, researchers can share or access anonymized data using a managed access process. To access anonymized individual patient-level data (IPD) arising from this project, users complete the Vivli data request form and sign the Vivli Data Use Agreement, which limits subsequent use to the terms of the approved proposal and requires that users maintain data security, and refrain from any attempts to re-identify research participants or engage in unauthorized uses of the data. Vivli will then make the data available via secure download. Researchers have a requirement to publish their findings as part of the Data Use Agreement and once the project is complete, must confirm that the original data and documents have been destroyed.
URL: https://vivli.org/